# **Cover Page**

Release Date: August 26, 2023

ClinicalTrials.gov ID: NCT03348670

Unique Protocol ID: IND 168800 to be IND EXEMPT

Brief Title: Pharmacogenomics IND EXEMPT SNP Clinical Study - Abiraterone and

Single Nucleotide Polymorphisms (Drugs-SNPs)

Official Title: Explore the Relationship Between Single Nucleotide Polymorphisms and

Abiraterone Response and Toxicity in Patients with Prostate Cancer.

**Secondary IDs:** FWA00015357 [Registry ID: HHS, Human Protections Administrator]

IRB00009424 [Registry ID: HHS, IRB] IORG0007849 [Registry ID: HHS, IORG]

NPI - 1831468511 [Registry ID: HHS, Health Care Provider Individual] NPI - 1023387701 [Registry ID: HHS, Health Care Provider Organization]

IND 168800 [Registry ID: FDA IND EXEMPT]

# **Contents**

| <b>21</b> C | CFR §312.23 (a)(3) | 2 |
|---|---|---|
| (3) | 3) Introductory statement and general investigational plan. | 2 |
| The | General Investigational plan [21 CFR 312.23(a)(3)] | 5 |
| > | Criteria: | 5 |
| > | Inclusion Criteria: | 5 |
| > | Exclusion Criteria: | 6 |
| The expected accrual populations: | | |
| Th | he primary efficacy and safety endpoints: | 6 |
| Th | he dose range (The statistical table): | 6 |
| Th | he analysis plans (The statistical analysis plan): | 7 |
| Th | he potential limitations of my proposed clinical trial: | 8 |
| Re | eference: | 8 |
| Rea | uest FDA approve IND 168800 to be IND EXEMPT SNP clinical trial NCT03348670: | 9 |

I think that my clinical study (NCT03348670) meets all of the requirements for exemption from the IND regulations [21 CFR 312.2(b)] and, therefore, an IND is not required to conduct my clinical investigation. The IND regulations [21 CFR 312.2(b)] state that my clinical investigation of oncology drug product (Abiraterone Tablet) that is lawfully marketed in the United States is exempt from the requirements for an IND, also is exempt from the requirements of this part (i.e., 21 CFR Part 312); i.e., my clinical investigation is exempt from all requirements in whole 21 CFR Part 312. My clinical investigation (NCT03348670) is not intended to be reported to FDA as a well-controlled study in support of a new indication for use, nor intended to be used to support any other significant change in the labeling for my oncology drug (Abiraterone Tablet). My investigation is not intended to support a significant change in the advertising for a prescription drug product; does not involve a change in route of administration, dosage level, or patient population, or other factor that significantly increases the risks (or decreases the acceptability of risks) associated with use of the drug product; is conducted in compliance with the requirements for institutional review (21 CFR Part 56) and informed consent (21 CFR Part 50); is conducted in compliance with the requirements of 21 CFR 312.7, i.e., the drug may not be represented as safe or effective for the purposes for which it is under investigation, nor may it be commercially distributed or sold. 21 CFR 312.2(b)(5) exempts from the IND requirements my clinical investigation that involves use of a placebo, and investigation does not otherwise require submission of an IND. My IND 168800 should be IND EXEMPT. The IND EXEMPT SNP clinical trial NCT03348670 will explore the relationship between single nucleotide polymorphisms and abiraterone response and toxicity in patients with prostate cancer. I request to initiate and conduct IND EXEMPT SNP clinical trial NCT03348670 based on IND 168800 to be IND EXEMPT.

# 21 CFR 312.2(b)(1)(iv)

### Statement

I write the <u>statement</u> with respect to each clinical study involving human subjects that it either will be conducted in compliance with the institutional review board regulations in part 56 or will not be subject to the regulations under §56.104 or §56.105; and that it either will be conducted in compliance with the informed consent regulations in part 50 or will not be subject to the regulations under §50.23 and §50.24.

## 21 CFR §312.23 (a)(3)

- (3) Introductory statement and general investigational plan.
- (i) A brief introductory statement giving the name of the drug and all active ingredients, the drug's pharmacological class, the structural formula of the drug (if known), the formulation of the dosage form(s) to be used, the route of administration, and the broad objectives and planned duration of the proposed clinical investigation(s).

The names of the drugs and all active ingredients:

NDC: 57894-195-06 (ZYTIGA - abiraterone acetate tablet, film coated) (NDA202379)

**NDC: 57894-150-12** (ZYTIGA - abiraterone acetate tablet) (NDA202379)

NDC: 0009-0045-01 (DELTASONE - prednisone tablet)

NDC:72974-120-01 (ORGOVYX- relugolix tablet, film coated) (NDA214621)

The drug's pharmacological class:

Antineoplastics (Oncology Drug)

The structural formula of the drug:

LABEL: ZYTIGA - Abiraterone Tablet (<a href="https://dailymed.nlm.nih.gov/dailymed">https://dailymed.nlm.nih.gov/dailymed</a>)

The formulation of the dosage form(s) to be used:

**Usual Approach Group** 

NDC: 57894-195-06 (ZYTIGA - abiraterone acetate tablet, film coated) ---

--- (2 x 500 mg tablets orally once daily) (12 weeks)

NDC: 0009-0045-01 (DELTASONE - Prednisone tablet) (5 mg orally twice daily) (12 weeks)

NDC:72974-120-01 (ORGOVYX - relugolix tablet, film coated) ---

--- (360 mg orally first day --- 120 mg orally once daily) (12 weeks)

Study Approach Group

NDC: 57894-150-12 (ZYTIGA - abiraterone acetate tablet) ---

--- (4 x 250 mg tablets orally once daily) (12 weeks)

NDC: 0009-0045-01 (DELTASONE - prednisone tablet) (5 mg orally once daily) (12 weeks)

NDC:72974-120-01 (ORGOVYX - relugolix tablet, film coated) ---

--- (360 mg orally first day --- 120 mg orally once daily) (12 weeks)

The route of administration:

Usual Approach Group: Oral Administration = OS

Study Approach Group: Oral Administration = OS

The broad objectives of my proposed clinical investigation:

Explore the relationship between single nucleotide polymorphisms and abiraterone response and toxicity in patients with prostate cancer.

The planned duration of my proposed clinical investigation:

90 days -- Phase 2 IND EXEMPT SNP Oncology Clinical Investigation NCT03348670

(ii) A brief summary of previous human experience with the drug, with reference to other IND's if pertinent, and to investigational or marketing experience in other countries that may be relevant to the safety of the proposed clinical investigation(s).

LABEL: ZYTIGA - Abiraterone Tablet (https://dailymed.nlm.nih.gov/dailymed)

(iii) If the drug has been withdrawn from investigation or marketing in any country for any reason related to safety or effectiveness, identification of the country(ies) where the drug was withdrawn and the reasons for the withdrawal.

The drug (ZYTIGA - Abiraterone Tablet) has <u>never</u> been withdrawn from investigation or marketing in any country for any reason related to safety or effectiveness.

(iv) A brief description of the overall plan for investigating the drug product for the following year. The plan should include the following: (a) The rationale for the drug or the research study: (b) the indication(s) to be studied: (c) the general approach to be followed in evaluating the drug: (d) the kinds of clinical trials to be conducted in the first year following the submission (if plans are not developed for the entire year, the sponsor should so indicate): (e) the estimated number of patients to be given the drug in those studies; and (f) any risks of particular severity or seriousness anticipated on the basis of the toxicological data in animals or prior studies in humans with the drug or related drugs.

# 90 days -- Phase 2 IND EXEMPT SNP Oncology Clinical Investigation NCT03348670

- (a) The rationale for the drug and the research study:
- The DNA gene chains are only formed by four types of nucleotides (Adenine = A; Thymine = T; Guanine = G; Cytosine = C). A single-nucleotide polymorphism (SNP) is a DNA sequence variation occurring a single nucleotide A, T, G, or C in a genome. Every SNP often has only two kinds of absolute different nucleotide composition forms, A<=>T or G<=>C. SNP is a dimorphic marker; if it is not A<=>T, it must be G<=>C; oppositely, if it is not G<=>C, it must be A<=>T. To almost all SNPs, every SNP is biallelic alleles, i.e., it only has two alleles as alternativa to all possible forms from all types of DNA nucleotides, A<=>T or G<=>C. Since every SNP should be a kind of ALL-OR-NONE gene mutation phenomenon, either it must have all, or it must have nothing all; this is almost same as the binary calculation of all computers, i.e., O<=>1 mode.
- ➢ Because SNP biallelic alleles genetics mode is almost same as the computer binary (0<=>1) calculation mode, SNP is the most suitable for high throughput analysing based on computer software. The first-selection analytical method to discover novel SNPs and to detect known SNPs is DNA precisely sequencing. Through high-throughput DNA precisely sequencing, high-throughput DNA sequence comparing, and high-throughput DNA chain genotyping, any one SNP will surely be found based on computer software analysing. Based on related computer software, any one drug target gene SNP will surely be found via drug target gene DNA strands' high-throughput DNA precisely sequencing, high-throughput DNA sequence comparing, and high-throughput DNA chain genotyping.
- The single-nucleotide polymorphisms (SNPs) are usually biallelic alleles and thus easily assayed by high-throughput DNA precisely sequencing. The now most cutting-edge DNA sequencing approach is the Oxford Nanopore DNA Sequencing uses electrophoresis to transport an unknown sample through an orifice of 10–9 meters in diameter. A nanopore system always contains an electrolytic solutions when a constant electric field is applied, an electric current can be observed in the system. The magnitude of the electric current density across a nanopore surface depends on the nanopore's dimensions and the composition of DNA or RNA that is occupying the nanopore. Sequencing is made possible because, when close enough to nanopores, samples cause characteristic changes in electric current density across nanopore surfaces. The total charge flowing through a nanopore channel is equal to

the surface integral of electric current density flux across the nanopore unit normal surfaces between times  $t_1$  and  $t_2$ . Oxford Nanopore DNA sequencing is referred to as "third generation" - "high-throughput" - "long-read" DNA sequencing technology. This approach is currently the world's most simple and efficient SNP detection and the highest accuracy rate of the method. In SNP clinical trial design, high-throughput DNA sequence comparing adopts the high-throughput genotyping based on above Oxford Nanopore DNA sequencing.

- ➤ Because every SNP has biallelic alleles ALL-OR-NONE characteristics, based on one drug target gene SNP analysing, every drug response test can only have one of two results, i.e. positive result (+) or negative result (-), i.e., every drug therapeutic effect (efficacy) test or every drug side effect (risk) test can only have one of two results, i.e. positive result (+) or negative result (-), so, the mechanism of pharmacology and toxicology of any drugs need never be guessed; the relationship between any drug target gene SNPs with any drug responses will be stable, and any drug target gene SNPs relating with any drug responses will surely be found. In SNP-pharmacogenomics clinical trials, if two double blind random separate groups' patients' drug target gene SNPs are the same; if the relationship between drug target gene SNPs and drug therapeutic effects are positive results (+), i.e. showing to have therapeutic effects, also if use these SNPs to define drug indication, this oncology drug chemotherapy efficacy can arrive higher than the 90% Effective Dose (ED90) level; if the relationship between drug target gene SNPs and drug side effects are negative results (-), i.e. showing to have no side effects, also if use these SNPs to define drug indication, this oncology drug chemotherapy risk can arrive lower than the 10% Lethal Dose (LD10) level.
- The classic oncology drug clinical trials must have placebo group, but the cancer patients in the placebo group will be equivalent to give up oncology drug treatments, so the placebo group cancer patients will surely die. But, because every SNP has biallelic alleles ALL-ORNONE characteristics, in same one SNP clinical trial, toward same one therapeutic effect or same one side effect, all two of double-blind random separate group patient drug target gene SNPs will be the same. Therefore, only need set up two double-blind random separate groups of patients, and then treat same one cancer with two different combination chemotherapies including same oncology drugs separately in two different treating groups; in these SNP-pharmacogenomics clinical trials, the placebo group will surely be avoided. Like as this, even in the SNP clinical trial stage, also can rescue much many cancer patients' lives.
- This clinical project's success means that the cancer organ system limitation of oncology drug chemotherapy will be broken-through, meanwhile, the cancer patient population who can use specific one oncology drug will be expanded. Because based on SNP biallelic alleles ALL-OR-NONE characteristics, if the same Oncology Drug Therapeutic Effect Target Gene SNP is detected in different cancers, when using the same drug, any kinds of cancers having the same drug therapeutic effect target gene SNP will have same therapeutic effect; so, any kinds of cancers having the same drug therapeutic effect target gene SNP will be suitable for using the same drug to treat.
  - (b) the indication(s) to be studied -- follow up Abiraterone Tablet DAILYMED Label:
  - LABEL: ZYTIGA Abiraterone Tablet (DAILYMED: <a href="https://dailymed.nlm.nih.gov">https://dailymed.nlm.nih.gov</a>)
  - Explore the relationship between single nucleotide polymorphisms and abiraterone response and toxicity in patients with prostate cancer.
  - (c) the general approach to be followed in evaluating the drug:
  - The usual approach to be followed in evaluating the drug (Abiraterone)
  - > The study approach to be followed in evaluating the drug (Abiraterone)

(d) the kinds of clinical trials to be conducted in the first year following the submission (if plans are not developed for the entire year, the sponsor should so indicate):

# 90 days -- Phase 2 IND EXEMPT SNP Oncology Clinical Trial NCT03348670

- (e) the estimated number of patients to be given the drug in those studies; ...
- The usual approach group: 300 patients with Prostate Cancer (PC)
- The study approach group: 300 patients with Prostate Cancer (PC)
- (f) any risks of particular severity or seriousness anticipated on the basis of the toxicological data in animals or prior studies in humans with the drug and related drugs.
  - LABEL: ZYTIGA Abiraterone Tablet (DailyMed: <a href="https://dailymed.nlm.nih.gov">https://dailymed.nlm.nih.gov</a>)
  - LABEL: DELTASONE prednisone tablet (DailyMed: <a href="https://dailymed.nlm.nih.gov">https://dailymed.nlm.nih.gov</a>)
  - LABEL: ORGOVYX relugolix tablet, film coated (DailyMed: <a href="https://dailymed.nlm.nih.gov">https://dailymed.nlm.nih.gov</a>)

# The General Investigational plan [21 CFR 312.23(a)(3)]

The study patients of **Prostate Cancer (PC)** will treat with abiraterone <u>without</u> prostate resection and follow up the <u>standard of care treatment with drug therapy</u> in the Abiraterone Tablet DAILYMED Label i.e., Recommended Dose for <u>Prostate Cancer (PC)</u> i.e., Abiraterone Tablet, DAILYMED in combination with other approved chemotherapeutic agents as first line treatment in patients with prostate cancer.

- > Criteria:
- ♦ Recruit 600 patients of **Prostate Cancer (PC)** without prostate resection.
- ♦ The 600 Prostate Cancer (PC) patients are randomly separated into 2 groups via computer.
- The usual approach randomization double-blinding active treatment concurrent control group:
- ✓ NDC: 57894-195-06 (ZYTIGA abiraterone acetate tablet, film coated) ---
  - --- (2 x 500 mg tablets orally once daily) (12 weeks)
- ✓ NDC: 0009-0045-01 (DELTASONE Prednisone tablet) (5 mg orally twice daily) (12 weeks)
- ✓ NDC:72974-120-01 (ORGOVYX- relugolix tablet, film coated) ---
  - --- (360 mg orally first day --- 120 mg orally once daily) (12 weeks)
- **♦** The study approach randomization double-blinding active treatment concurrent control group:
- ✓ NDC: 57894-150-12 (ZYTIGA abiraterone acetate tablet) -- (4 x 250 mg tablets orally once daily) (12 weeks)
- ✓ NDC: 0009-0045-01 (DELTASONE Prednisone tablet) (5 mg orally once daily) (12 weeks)
- ✓ NDC: 72974-120-01 (ORGOVYX- relugolix tablet, film coated) ---
  - --- (360 mg orally first day --- 120 mg orally once daily) (12 weeks)
- ♦ Every prostate cancer patient will receive peripheral blood-drawing.
- ♦ Keep storing all peripheral blood.
- ♦ All participating patients image test at least one time per month.
- ♦ All participating patients will need urine tests every week while they are taking oncology drugs.
- ♦ All participating patients will need blood tests every week while they are taking oncology drugs.
- ♦ Sequence precisely each target gene DNA whole chain in peripheral blood like as following: CYP17, SULT2A1, GnRH-R, CYP3A (CYP3A4, CYP3A5, CYP3A7, CYP3A43), CYP2C8.
- ♦ If any participating patients have serious side effects, they will be stopped the research.
- ♦ If any participating patients have no therapeutic effects, they will be stopped the research.
- > Inclusion Criteria:
- 1. Clinical diagnosis of Prostate Cancer (PC) without prostate resection
- 2. Random and double blind

- 3. Measurable disease
- 4. Adequate organ functions
- 5. Adequate performance status
- 6. Age 22 years old and over
- 7. Receive blood-drawing.
- 8. Sign an informed consent form.

#### Exclusion Criteria:

- 1. Treatment with other anti-cancer therapies and the therapies cannot be stopped currently.
- 2. The patients with other serious inter-current illness or infectious diseases
- 3. Have more than one different kind of cancer at the same time
- 4. Serious Allergy Tendency
- 5. Serious Bleed Tendency
- 6. Serious Risks or Serious Adverse Events of the drug product
- 7. The prohibition of the drug product
- 8. The participating patients have serious side effects.
- 9. The participating patients have no therapeutic effects.

### The expected accrual populations:

- ♦ Recruit 600 patients with Prostate Cancer (PC) without prostate resection.
- ♦ The 600 PC patients are randomly separated into 2 groups via computer.
- ♦ The usual approach group is 300 PC patients.
- ♦ The study approach group is 300 PC patients.
- → Every PC patient will receive peripheral blood-drawing.
- ♦ Keep storing all peripheral blood.

### The primary efficacy and safety endpoints:

- After clinical diagnosis of prostate cancer (PC), through usual approach combined chemotherapy or study approach combined chemotherapy, in 90-days Phase 2 IND EXEMPT SNP Oncology Clinical Trial, there should **not** be cancer growth or cancer metastasis.
- If appear cancer growth or cancer metastasis, stop these patients' trial.
- If appear serious side effects or serious adverse reactions, stop these patients' trial.

### The dose range (The statistical table):

- ♦ The usual approach randomization double-blinding active treatment concurrent control group:
- ✓ ZYTIGA abiraterone acetate tablet, film coated --- 2 x 500 mg tablets orally once daily (12 weeks)
- ✓ DELTASONE Prednisone tablet --- 5 mg orally twice daily (12 weeks)
- ✓ ORGOVYX- relugolix tablet, film coated --- 360 mg orally first day 120 mg orally once daily (12 weeks)

| Drug Names | Targets in Peripheral Blood |
|---|---|
| Abiraterone Tablet | CYP17<br>CYP3A4<br>SULT2A1 |
| Relugolix Tablet | GnRH Receptor<br>CYP3A (CYP3A4, CYP3A5, CYP3A7, CYP3A43)<br>CYP2C8 |

- ♦ The study approach randomization double-blinding active treatment concurrent control group:
- ✓ ZYTIGA abiraterone acetate tablet, film coated --- 2 x 500 mg tablets orally once daily (12 weeks)
- ✓ DELTASONE Prednisone tablet --- 5 mg orally once daily (12 weeks)
- ✓ ORGOVYX- relugolix tablet, film coated --- 360 mg orally first day 120 mg orally once daily (12 weeks)

| Drug Names | Targets in Peripheral Blood |
|---|---|
| Abiraterone Tablet | CYP17<br>CYP3A4<br>SULT2A1 |
| Relugolix Tablet | GnRH Receptor<br>CYP3A (CYP3A4, CYP3A5, CYP3A7, CYP3A43)<br>CYP2C8 |

### The analysis plans (The statistical analysis plan):

- ♦ 600 PC patients will test peripheral blood DNA.
- ✓ Every PC patient will receive testing CYP17 Gene SNPs in peripheral blood DNA.
- ✓ Every PC patient will receive testing SULT2A1 Gene SNPs in peripheral blood DNA.
- ✓ Every PC patient will receive testing GnRH-R Gene SNPs in peripheral blood DNA.
- ✓ Every PC patient will receive testing CYP3A (CYP3A4) Gene SNPs in peripheral blood DNA.
- ✓ Every PC patient will receive testing CYP3A (CYP3A5) Gene SNPs in peripheral blood DNA.
- Every PC patient will receive testing CYP3A (CYP3A7) Gene SNPs in peripheral blood DNA.
- ✓ Every PC patient will receive testing CYP3A (CYP3A43) Gene SNPs in peripheral blood DNA.
- ✓ Every PC patient will receive testing CYP2C8 Gene SNPs in peripheral blood DNA.
- ♦ Sequence precisely CYP17, SULT2A1, GnRH-R, CYP3A (CYP3A4, CYP3A5, CYP3A7, CYP3A43), CYP2C8 gene DNA whole chain in peripheral blood.
- ✓ Find every single nucleotide gene mutation site in every oncology drug target gene DNA whole chain.
- ✓ Find every single nucleotide gene mutation site in CYP17, SULT2A1, GnRH-R, CYP3A (CYP3A4, CYP3A5, CYP3A7, CYP3A43), CYP2C8 gene DNA whole chain.
- ♦ If one single nucleotide gene mutation site appears ratio more than 1% in 600 PC patients, this is SNP.
- ✓ Calculate CYP17 Gene SNPs in peripheral blood DNA in 600 PC patients.
- ✓ Calculate SULT2A1 Gene SNPs in peripheral blood DNA in 600 PC patients.
- ✓ Calculate GnRH-R Gene SNPs in peripheral blood DNA in 600 PC patients.
- ✓ Calculate CYP3A (CYP3A4) Gene SNPs in peripheral blood DNA in 600 PC patients.
- ✓ Calculate CYP3A (CYP3A5) Gene SNPs in peripheral blood DNA in 600 PC patients.
- ✓ Calculate CYP3A (CYP3A7) Gene SNPs in peripheral blood DNA in 600 PC patients.
- ✓ Calculate CYP3A (CYP3A43) Gene SNPs in peripheral blood DNA in 600 PC patients.
- ✓ Calculate CYP2C8 Gene SNPs in peripheral blood DNA in 600 PC patients.
- ❖ If the peripheral blood samples of the usual approach group have the same oncology drug target gene SNP as the peripheral blood samples of the study approach group, the relationship between this oncology drug target gene SNP and this oncology drug efficacy can be confirmed, i.e., this oncology drug target gene SNP is relating to this oncology drug efficacy.
- ♦ If the peripheral blood samples of the usual approach group have the same CYP17 gene SNP as the peripheral blood samples of the study approach group, the relationship between this CYP17 gene SNP and this ABIRATERONE oncology drug efficacy can be confirmed, i.e., this CYP17 gene SNP is relating to this ABIRATERONE oncology drug efficacy.
- ♦ If the peripheral blood samples of the usual approach group have the same GnRH-R gene SNP as the peripheral blood samples of the study approach group, the relationship between this GnRH-R gene SNP and this RELUGOLIX oncology drug efficacy can be confirmed, i.e., this GnRH-R gene SNP is relating to this RELUGOLIX oncology drug efficacy.

| Target Gene SNP in peripheral blood of Usual Approach Group of an PC patient | Target Gene SNP in peripheral blood of Study Approach Group of an PC patient | Comparing Results |
|---|---|---|
| CYP17 gene SNP | CYP17 gene SNP | Same |
| This CYP17 gene SNP is related to the ABIRATERONE drug efficacy. | | |
| Target Gene SNP in peripheral blood of Usual Approach Group of an PC patient | Target Gene SNP in peripheral blood of Study Approach Group of an PC patient | Comparing Results |
| GnRH-R gene SNP | GnRH-R gene SNP | Same |
| This GnRH-R gene SNP is related to the RELUGOLIX drug efficacy. | | |

- ❖ If the peripheral blood samples of the usual approach group have the same oncology drug target gene SNP as the peripheral blood samples of the study approach group, the relationship between this oncology drug target gene SNP and this oncology drug risk can be confirmed, i.e., this oncology drug target gene SNP is relating to this oncology drug risk.
- ❖ If the peripheral blood samples of the usual approach group have the same CYP3A4 gene SNP as the peripheral blood samples of the study approach group, the relationship between this SULT2A1 gene SNP and this ABIRATERONE drug risk can be confirmed, i.e., this SULT2A1 gene SNP is relating to this ABIRATERONE drug risk.

| Target Gene SNP in Peripheral Blood of Usual<br>Approach Group of an PC patient | Target Gene SNP in Peripheral Blood of Study<br>Approach Group of an PC patient | Comparing Results |
|---|---|---|
| SULT2A1 gene SNP | SULT2A1 gene SNP | Same |
| CYP3A (CYP3A4) gene SNP | CYP3A (CYP3A4) gene SNP | Different |
| CYP3A (CYP3A5) gene SNP | CYP3A (CYP3A5) gene SNP | Different |
| CYP3A (CYP3A7) gene SNP | CYP3A (CYP3A7) gene SNP | Different |
| CYP3A (CYP3A43) gene SNP | CYP3A (CYP3A43) gene SNP | Different |
| CYP2C8 gene SNP | CYP2C8 gene SNP | Different |
| This SULT2A1 Gene SNP is related to the ABIRATERONE drug risk. | | |

# The potential limitations of my proposed clinical trial:

The study patients will be treated the **Prostate Cancer (PC)** with ABIRATERONE <u>without</u> prostate resection. The IND EXEMPT SNP investigation will follow up the standard of care treatment with drug therapy in the ZYTIGA - Abiraterone Tablet DAILYMED Label.

I (Han Xu, M.D., Ph.D. i.e., Sponsor i.e., Sponsor-Investigator) as IRB Chair of our IRB (IRB00009424) will only organize the IRB meeting but give up my voting power in the IRB determination, when I conduct my clinical investigation (NCT03348670).

#### Reference:

- LABEL: ZYTIGA Abiraterone Tablet (DAILYMED: https://dailymed.nlm.nih.gov)
- > LABEL: DELTASONE Prednisone tablet (DAILYMED: https://dailymed.nlm.nih.gov)
- LABEL: ORGOVYX relugolix tablet, film coated (DAILYMED: <a href="https://dailymed.nlm.nih.gov">https://dailymed.nlm.nih.gov</a>)

## Request FDA approve IND 168800 to be IND EXEMPT SNP clinical trial NCT03348670:

My clinical study (NCT03348670) meets all of the requirements for exemption from the IND regulations and, therefore, an IND is not required to conduct my clinical investigation; i.e., my clinical investigation of oncology drug product (Abiraterone Tablet) that is lawfully marketed in the United States is exempt from the requirements for an IND, also is exempt from the requirements of this part (i.e., 21 CFR Part 312); i.e., my clinical investigation is exempt from the requirements of investigator in whole 21 CFR Part 312: i.e., my clinical investigation is exempt from the requirements of 21 CFR §312.305 (c)(1) and 21 CFR §312.305 (c)(3). Although I am not a licensed physician, I still can be a qualified investigator for my IND EXEMPT SNP oncology drug clinical investigation. In my APCR documents, Han Xu, M.D., Ph.D., FAPCR had been defined as PI (Principal Investigator) in clinical trials. In my document ClinicalTrials.gov ID: NCT03348670, I (Han Xu, M.D., Ph.D., FAPCR) am defined as Responsible Party (Sponsor-Investigator) and Study Principal Investigator [Principal Investigator (PI)]. So, Han Xu, M.D., Ph.D. must be the sponsor-investigator (S-I) of my clinical trial. So, I (Han Xu, M.D., Ph.D. i.e., Sponsor i.e., Sponsor-Investigator) can both initiate and conduct, alone or with others, my clinical investigation (NCT03348670).

My clinical investigation (NCT03348670) is not intended to be reported to FDA as a well-controlled study in support of a new indication for use, nor intended to be used to support any other significant change in the labeling for my oncology drug (Abiraterone Tablet). My investigation is not intended to support a significant change in the advertising for a prescription drug product; does not involve a change in route of administration, dosage level, or patient population, or other factor that significantly increases the risks (or decreases the acceptability of risks) associated with use of the drug product; is conducted in compliance with the requirements for institutional review (21 CFR Part 56) and informed consent (21 CFR Part 50); is conducted in compliance with the requirements of 21 CFR 312.7, i.e., the drug may not be represented as safe or effective for the purposes for which it is under investigation, nor may it be commercially distributed or sold. 21 CFR 312.2(b)(5) exempts from the IND requirements my clinical investigation that involves use of a placebo, and investigation does not otherwise require submission of an IND. My IND 168800 should be IND EXEMPT. The IND EXEMPT SNP clinical trial NCT03348670 will explore the relationship between single nucleotide polymorphisms and abiraterone response and toxicity in patients with prostate cancer. I am requesting FDA approve my IND 168800 to be IND EXEMPT SNP clinical trial NCT03348670 via this pre-IND meeting with Written response only -- WRO by email.

### 21 CFR 312.2(b)(1)(iv)

The investigation is conducted in compliance with the requirements for institutional review set forth in part 56 and with the requirements for informed consent set forth in part 50.

### Statement

I write the <u>statement</u> with respect to each clinical study involving human subjects that it either will be conducted in compliance with the institutional review board regulations in part 56 or will not be subject to the regulations under §56.104 or §56.105; and that it either will be conducted in compliance with the informed consent regulations in part 50 or will not be subject to the regulations under §50.23 and §50.24.

According to 21 CFR 56.102(g), Institutional Review Board (IRB) can approve the initiation of, and can conduct periodic review of, biomedical research involving human subjects.

According to 21 CFR 56.102(m), IRB approval means the determination of our IRB (IRB00009424) that my clinical investigation (NCT03348670) has been reviewed and may be conducted at our institution (Medicine Invention Design Incorporation) within the constraints set forth by our IRB (IRB00009424) and by other institutional and Federal requirements.

I (Han Xu, M.D., Ph.D. i.e., Sponsor i.e., Sponsor-Investigator) as IRB Chair of our IRB (IRB00009424) will only organize the IRB meeting but give up my voting power in the determination of IRB, when I conduct my clinical investigation (NCT03348670).